CLINICAL TRIAL: NCT02484911
Title: Aprepitant ,Olanzapine,Palonosetron and Dexamethasone for the Prevention of Chemotherapy-induced Nausea and Vomiting---A Randomized Single Center Phase III Trial
Brief Title: Aprepitant ,Olanzapine,Palonosetron and Dexamethasone for the Prevention of Chemotherapy-induced Nausea and Vomiting
Acronym: AOPDPCINV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GHYDZ-1225
Record Dates: First submitted 2015-06-22; First posted 2015-06-30 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2016-06

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: chemotherapy nausea vomiting
MeSH Terms: conditions — Vomiting | interventions — Olanzapine; Aprepitant; Palonosetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olanzapine regimen (Experimental): Olanzapine in combination with aprepitant ,palonosetron and dexamethasone.
  Interventions: Drug: Olanzapine; Drug: Aprepitant; Drug: Palonosetron; Drug: Dexamethasone
- Control regimen (Other): Aprepitant in combination with palonosetron and dexamethasone
  Interventions: Drug: Aprepitant; Drug: Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Olanzapine — 5mg,twice a day orally on day 1 to day 4
  Arms: Olanzapine regimen
Drug: Aprepitant — 125 mg capsule per oral, 1 hour before chemotherapy on day 1, 80 mg capsule daily in the morning during days 2 to 3.
Drug: Palonosetron — 0.25mg IV 30-60min before chemotherapy on day 1
Drug: Dexamethasone — 6mg IV on day 1 ，3.75mg IV on day 2 to 4

SUMMARY:
The purpose of the study is to mainly evaluate the efficacy and safety of aprepitant in combination with olanzapine ,palonosetron and dexamethasone for the prevention of chemotherapy-induced nausea and vomiting (CINV) in patients receiving highly or moderately emetogenic chemotherapy.

DETAILED DESCRIPTION:
Eligible patients will be randomized to receive different antiemetic regimens . In the experimental group,patients will receive aprepitant,olanzapine ,palonosetron and dexamethasone .In the other group,patients will accept the same dose of aprepitant ,palonosetron and dexamethasone .During the treatment, any grade of nausea and vomiting should be recorded in order to evaluate the complete response rate of CINV,nausea patients will be measured by a visual analogue scale (VAS) ,other adverse events should be recorded as well.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Histologically or cytologically confirmed malignant disease
3. Accept chemotherapy for the first time
4. Patients who will receive high emetogenic cancer chemotherapy (HEC) (cisplatin>=70mg/m2,adriamycin in combination with cyclophosphamide ,cyclophosphamide>=1500mg/m2,adriamycin>60mg/m2,epirubicin>90mg/m2,dacarbazine，ifosfamide>=2g/m2) or moderate emetogenic chemotherapy cancer (carboplatin>=300mg/m2,cyclophosphamide>=600-1000mg/m2,adriamycin>50mg/m2)
5. Written informed consent

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Uncontrolled psychosis history
3. Inability or unwillingness to understand or cooperate with study procedures
4. Central nervous system tumors primary or secondary
5. Concurrent abdominal radiotherapy
6. History of uncontrolled diabetes mellitus
7. Patients of prostatic hyperplasia ，paralytic ileus，narrow feet glaucoma.
8. Known cardiac arrhythmia, uncontrolled congestive heart failure ,or acute myocardial infarction with the previous six month
9. Pre-existing nausea or vomiting
10. Inadequate hematological function and abnormal liver and renal function.
11. History of sensitivity to olanzapine
12. Concurrent application of quinolone antibiotic therapy
13. Treatment with another antipsychotic agent such as risperidone,quetiapine, clozapine,phenothiazine,or butyrophenone for 30 days prior to or during the chemotherapy.
14. Cytochrome P450 3A4 substrates within 7 days (terfenadine, cisapride, astemizole, pimozide)
15. Concurrent application of systemic corticosteroids
16. Active infection or gastrointestinal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daxin Zhang, MD, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

REFERENCES:
- [Background] Andrews PL, Naylor RJ, Joss RA. Neuropharmacology of emesis and its relevance to anti-emetic therapy. Consensus and controversies. Support Care Cancer. 1998 May;6(3):197-203. doi: 10.1007/s005200050154. PMID 9629870
- [Background] Matsuki N, Torii Y, Saito H. Effects of iron and deferoxamine on cisplatin-induced emesis: further evidence for the role of free radicals. Eur J Pharmacol. 1993 Dec 1;248(4):329-31. doi: 10.1016/0926-6917(93)90008-e. PMID 8181539
- [Background] Tattersall FD, Rycroft W, Cumberbatch M, Mason G, Tye S, Williamson DJ, Hale JJ, Mills SG, Finke PE, MacCoss M, Sadowski S, Ber E, Cascieri M, Hill RG, MacIntyre DE, Hargreaves RJ. The novel NK1 receptor antagonist MK-0869 (L-754,030) and its water soluble phosphoryl prodrug, L-758,298, inhibit acute and delayed cisplatin-induced emesis in ferrets. Neuropharmacology. 2000 Feb 14;39(4):652-63. doi: 10.1016/s0028-3908(99)00172-0. PMID 10728886
- [Result] Hesketh PJ, Van Belle S, Aapro M, Tattersall FD, Naylor RJ, Hargreaves R, Carides AD, Evans JK, Horgan KJ. Differential involvement of neurotransmitters through the time course of cisplatin-induced emesis as revealed by therapy with specific receptor antagonists. Eur J Cancer. 2003 May;39(8):1074-80. doi: 10.1016/s0959-8049(02)00674-3. PMID 12736106
- [Result] Grunberg SM, Hesketh PJ. Control of chemotherapy-induced emesis. N Engl J Med. 1993 Dec 9;329(24):1790-6. doi: 10.1056/NEJM199312093292408. PMID 8232489
- [Result] Grunberg SM, Slusher B, Rugo HS. Emerging treatments in chemotherapy-induced nausea and vomiting. Clin Adv Hematol Oncol. 2013 Feb;11(2 Suppl 1):1-18; quiz 2 p following 18. PMID 23598819
- [Result] Diemunsch P, Grelot L. Potential of substance P antagonists as antiemetics. Drugs. 2000 Sep;60(3):533-46. doi: 10.2165/00003495-200060030-00002. PMID 11030465
- [Result] Gao HF, Liang Y, Zhou NN, Zhang DS, Wu HY. Aprepitant plus palonosetron and dexamethasone for prevention of chemotherapy-induced nausea and vomiting in patients receiving multiple-day cisplatin chemotherapy. Intern Med J. 2013 Jan;43(1):73-6. doi: 10.1111/j.1445-5994.2011.02637.x. PMID 22141732
- [Result] Tan L, Liu J, Liu X, Chen J, Yan Z, Yang H, Zhang D. Clinical research of Olanzapine for prevention of chemotherapy-induced nausea and vomiting. J Exp Clin Cancer Res. 2009 Sep 23;28(1):131. doi: 10.1186/1756-9966-28-131. PMID 19775450
- [Result] Navari RM, Gray SE, Kerr AC. Olanzapine versus aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a randomized phase III trial. J Support Oncol. 2011 Sep-Oct;9(5):188-95. doi: 10.1016/j.suponc.2011.05.002. Epub 2011 Sep 24. PMID 22024310
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Differential+involvement+of+neurotransmitters+through+the+time+course+of+cisplatin-induced+emesis+as+revealed+by+therapy+with+specific+receptor+antagonists
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/8232489
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Effects+of+iron+and+deferoxamine+on+cisplatin-induced+emesis%3A+further+evidence+for+the+role+of+free+radicals
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23598819
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Diemunsch+P%2C+Grelot+L.+et+al.+Potential+of+substance+P+antagonists+as+antiemetics
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=The+novel+NK1+receptor+antagonist+MK-0869+(L-754%2C030)+and+its+water+soluble+phosphoryl+prodrug%2C+L-758%2C298%2C+inhibit+acute+and+delayed+cisplatin-induced+emesis+in+ferrets.+Neuropharmacology.
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22141732
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19775450
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22024310

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olanzapine Regimen | Control Regimen
Started | 60 | 60
Completed | 56 | 58
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine Regimen | Control Regimen | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 49 | 96
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (9.55) | 52.98 (10.81) | 54.18 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 23 | 21 | 44
Region of Enrollment [Number; unit: participants]
  China | 56 | 56 | 114
History of drinking [Number; unit: participants]
  YES | 15 | 9 | 24
  NO | 41 | 49 | 90

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Receiving HEC With Complete Response in Overall Phase
Description: Overall phase was defined as 0 to 120 hours following initiation of chemotherapy.
  Complete response was defined as no vomiting with no rescue therapy.
Time Frame: 0 to 120 hours
Population: FAS (full analysis set) patient population was used for all efficacy evaluations and included patients who (1) received High Emetogenic Chemotherapy (HEC), (2) took a dose of study drug, and (3) completed treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Olanzapine Regimen: Day 1:Olanzapine: 5mg twice po Aprepitant :125mg one hour po before chemotherapy Palonosetron :0.25mg IV 30-60min before chemotherapy Dexamethasone: 6mg IV Day 2-Day3: Olanzapine: 5mg twice Aprepitant:80mg po Dexamethasone: 3.75mg IV Day4: Olanzapine 5mg twice po Dexamethasone: 3.75mg IV
- Control Regimen: Day1： Aprepitant :125mg one hour before chemotherapy po, Palonosetron :0.25mg IV 30-60min before chemotherapy Dexamethasone: 6mg IV
  Day2-Day3:
  Olanzapine: 5mg twice Aprepitant:80mg po Dexamethasone: 3.75mg IV
  Day4:
  Olanzapine 5mg twice po Dexamethasone: 3.75mg IV
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 20 | 17
Participants | 20 | 15
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.397, Chi-squared

2. Primary Outcome: Proportion of Participants Receiving MEC With Complete Response in Overall Phase
Description: as for outcome 1
Time Frame: 0 to 120 hours
Population: FAS (full analysis set) patient population was used for all efficacy evaluations and included patients who (1) received Moderate Emetogenic Chemotherapy (MEC), (2) took a dose of study drug, and (3) completed treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 36 | 41
Participants | 36 | 40
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 1.0, Chi-squared

3. Secondary Outcome: Proportion of Participants Receiving HEC With Complete Response in the Acute Phase
Description: Acute phase was defined as 0 to 24 hours following initiation of chemotherapy. Complete response was defined as no vomiting with no rescue therapy.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 20 | 17
Participants | 20 | 17

4. Secondary Outcome: Proportion of Participants Receiving HEC With Complete Response in the Delayed Phase
Description: Delayed phase was defined as 24 to 120 hours following initiation of chemotherapy.
  Complete response was defined as no vomiting with no rescue therapy.
Time Frame: 24 to 120 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Aprepitant Regimen: Day1： Aprepitant :125mg one hour before chemotherapy po, Palonosetron :0.25mg IV 30-60min before chemotherapy Dexamethasone: 6mg IV
  Day2-Day3:
  Olanzapine: 5mg twice Aprepitant:80mg po Dexamethasone: 3.75mg IV
  Day4:
  Olanzapine 5mg twice po Dexamethasone: 3.75mg IV
Arm/Group | Olanzapine Regimen | Aprepitant Regimen
Number analyzed (Participants) | 20 | 17
Participants | 20 | 15
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Aprepitant Regimen; Test type: Superiority or Other; p = 0.397, Chi-squared

5. Secondary Outcome: Proportion of Participants Receiving HEC With No Vomiting in the Overall Phase
Description: Overall phase was defined as 0 to 120 hours following initiation of chemotherapy.
  No vomiting was defined as no vomiting or retching or dry heaves (included participants who received rescue therapy).
Time Frame: 0 to 120 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 20 | 17
Participants | 17 | 6
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.02, Chi-squared

6. Secondary Outcome: Proportion of Participants Receiving HEC With No Vomiting in the Acute Phase
Description: Overall Phase was defined as 0 to 120 hours following initiation of chemotherapy.
  No vomiting was defined as no vomiting or retching or dry heaves (included participants who received rescue ）
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 20 | 17
Participants | 18 | 15
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 1.0, Chi-squared

7. Secondary Outcome: Proportion of Participants Receiving HEC With No Vomiting in the Delayed Phase
Description: Overall Phase was defined as 24 to 120 hours following initiation of chemotherapy.
  No vomiting was defined as no vomiting or retching or dry heaves (included participants who received rescue therapy).
Time Frame: 24 to 120 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 20 | 17
Participants | 17 | 7
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.005, Chi-squared

8. Secondary Outcome: Proportion of Participants Receiving MEC With Complete Response in the Acute Phase
Description: as for outcome 3
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 36 | 41
Participants | 36 | 41

9. Secondary Outcome: Proportion of Participants Receiving MEC With Complete Response in the Delayed Phase
Description: as for outcome 4
Time Frame: 24 to 120 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 36 | 41
Participants | 36 | 40
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 1.0, Chi-squared

10. Secondary Outcome: Proportion of Participants Receiving MEC With No Vomiting in the Overall Phase
Description: as for outcome 5
Time Frame: 0-120 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 36 | 41
Participants | 30 | 30
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.283, Chi-squared

11. Secondary Outcome: Proportion of Participants Receiving MEC With No Vomiting in the Acute Phase
Description: Overall Phase was defined as 0 to 24 hours following initiation of chemotherapy.
  No vomiting was defined as no vomiting or retching or dry heaves (included participants who received rescue therapy).
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 36 | 41
Participants | 35 | 40
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 1.0, Chi-squared

12. Secondary Outcome: Proportion of Participants Receiving MEC With No Vomiting in the Delayed Phase
Description: as for outcome 7
Time Frame: 24 to 120 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine Regimen | Control Regimen
Number analyzed (Participants) | 36 | 41
Participants | 30 | 31
Statistical Analysis 1: Comparison: Olanzapine Regimen vs Control Regimen; Test type: Superiority or Other; p = 0.246, Chi-squared

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 6, inclusive
Description: The Safety population consisted of all participants who received study drug. Participants are included in the treatment group based on the study drug they actually received
Arm/Group | Olanzapine Regimen | Control Regimen
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 21/56 | 14/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olanzapine Regimen (N=56) | Control Regimen (N=58)
Abdominal distension (Gastrointestinal disorders) | 4 | 5
Drowsiness (Nervous system disorders) | 11 | 0
Dizzy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 3
Fatigue (General disorders) | 0 | 2
dry mouth (General disorders) | 1 | 1
Oral ulcer (General disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes